CLINICAL TRIAL: NCT01614405
Title: Randomized Controlled Pilot Study of Highly Active Anti-Retroviral Therapy for Patients With Primary Biliary Cirrhosis
Brief Title: Highly Active Antiretroviral Therapy for Patients With Primary Biliary Cirrhosis
Acronym: HAART
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Protracted gastrointestinal symptoms were experienced by most patients who were subsequently found to be in the treatment arm on LPV/r. This observation resulted in cessation of enrolment and a decision not to continue the RCT
Sponsor: University of Alberta (Other)
Collaborators: Abbott (Industry); Gilead Sciences (Industry); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HAART Study
Record Dates: First submitted 2011-04-25; First posted 2012-06-07 (Estimated); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Primary Biliary Cirrhosis
Keywords: PBC
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Tenofovir; Emtricitabine; lopinavir-ritonavir drug combination; Lopinavir; Ritonavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Identical Placebo Tablets.
  Duration: 6 months therapy with blinded placebo followed by 6 months open label therapy (Truvada and Kaletra). Following, there is an option for an 18-month extension study.
  Interventions: Drug: Placebo
- TDF/FTC/LPV/r (Active Comparator): TDF/FTC/LPV/r
  One tablet of Truvada a day at standard dose of Tenofovir 300mg and Emtricitabine 200mg and four tablets of Kaletra once a day for a total dose of lopinavir 800mg and ritonavir 200mg for 6 months, or less if adverse events occur.
  Duration: 6 months of therapy with the option of open label for additional 18-month extension study.
  Interventions: Drug: TDF/FTC/LPV/r

INTERVENTIONS:
Drug: TDF/FTC/LPV/r — one tablet of Truvada a day at standard dose of Tenofovir 300mg and Emtricitabine 200mg and four tablets of Kaletra once a day for a total dose of lopinavir 800mg and ritonavir 200mg for 6 months or less if adverse events occur
  Other Names: Truvada; Tenofovir; Emtricitabine; Kaletra; lopinavir; ritonavir
  Arms: TDF/FTC/LPV/r
Drug: Placebo — 6 months therapy with blinded placebo followed by 6 months open label therapy with Kaletra and Truvada.
  Other Names: Truvada; Tenofovir; Emtricitabine; lopinavir; ritonavir
  Arms: Placebo

SUMMARY:
Patients with primary biliary cirrhosis (PBC) develop progressive liver disease and often require liver transplantation. The cause of disease is unknown. It is thought to occur as a result of an infection in subjects that are more susceptible to disease than others. The investigators found evidence of retrovirus infection in patients with primary biliary cirrhosis. The investigators found that most patients with PBC have evidence of viral infection. Since then the investigators have conducted clinical studies using anti-viral therapy. The investigators found that PBC patients treated with combination anti-retrovirus therapy experienced significant reversal of the disease process. However, the changes were not substantial and the investigators are now looking for better antiviral regimens. Now the investigators have found a mouse model with a similar virus infection that develops a similar biliary disease. Importantly, the investigators found that antiviral therapy blocks the development of the disease in this mouse. The investigators have used this model to find safer and more effective antiviral treatments for patients with PBC. The investigators have now found out that a combination of highly active antiretroviral therapy with Truvada and Kaletra stops disease in the mouse and plan to use this combination to see if it works in patients with PBC.

DETAILED DESCRIPTION:
6 months therapy with blinded Kaletra and Truvada vs. 6 months therapy with blinded placebo followed by 6 months open label therapy with Kaletra and Truvada

18 month extension study with open label Kaletra and Truvada in patients completing 6 months of therapy with Kaletra and Truvada with biochemical endpoint

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years old of either sex will be recruited for this study.
2. Elevated ALP after 6 months UDCA therapy ≥ 2 x upper limit of normal or abnormal bilirubin.
3. Positive serum AMA or Liver biopsy histology compatible with PBC.
4. Maintained on UDCA at a dose of 13-15 mg/kg for 6 or more months.
5. Patients must read and sign informed consent form

Exclusion Criteria:

1. Subjects with baseline AST or ALT > 5 x ULN.
2. Patients who have altered dose of any medications used to treat PBC (such as UDCA) or the use of colchicine, corticosteroids, azathioprine, chlorambucil, methotrexate, or D-penicillamine within the last 6 months.
3. Advanced liver disease or esophageal varices, INR > 1.2 (upper limit of normal), Albumin < 35 g/L (lower limit of normal), platelets < 120,000/mm3, Childs Pugh class B or C cirrhosis, presence of varices or previous variceal hemorrhage, spontaneous encephalopathy, ascites or need for liver transplantation.
4. Patients with a secondary diagnosis such as HIV, viral hepatitis, drug induced liver injury, extrahepatic biliary obstruction, primary sclerosing cholangitis, metabolic liver diseases or alcoholic liver disease Regular use of more than 30 g of alcohol per day in the last year. Clinically apparent pancreatitis or with a predicted survival of less than 3 years from malignant or other potentially life threatening disease.
5. An ultrasound showing a hepatic mass consistent with hepatocellular carcinoma within the last year in patients with cirrhosis.
6. Previous allergic reaction to study medications.
7. Creatinine clearance less than < 70 mL/min using the Cockcroft Gault equation:

   Creatinine clearance (mL/min) = (140 - age) x body wt (Kg) x 0.85 (if female)/serum creatinine in mol/l
8. Pregnancy or breast-feeding a child. Young sexually active patients not using contraception
9. Young sexually active patients not using contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-06; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Reduction of ALP to 1.67x ULN | The outcomes will be measured are from 12 to 24 weeks at the end of the study
normalization of bilirubin. | The outcomes will be measured are from 12 to 24 weeks at the end of the study

SECONDARY OUTCOMES:
Reduction of human betaretrovirus. | The outcomes will be measured are from 12 to 24 weeks in RCT; and 6 monthly to 2 years for the extension study
Symptoms with changes in PBC-40 | The outcomes will be measured are from 12 to 24 weeks in RCT; and 6 monthly to 2 years for the extension study
Changes in AMA and immunoglobulin levels | The outcomes will be measured are from 12 to 24 weeks in RCT; and 6 monthly to 2 years for the extension study
Biochemistry: GGT, AST and ALT | The outcomes will be measured are from 12 to 24 weeks in RCT; and 6 monthly to 2 years for the extension study
Histology in extension study | The outcomes will be measured are from 12 to 24 weeks in RCT; and 6 monthly to 2 years for the extension study

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Mason, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Schembri G, Schober P. Killing two birds with one stone. Lancet. 2011 Jan 1;377(9759):96. doi: 10.1016/S0140-6736(10)61343-8. No abstract available. PMID 21195252